CLINICAL TRIAL: NCT05558904
Title: Positron-Emission Tomography Detection of Sodium-Glucose Transport for Early Diagnosis of Lung Cancer
Brief Title: An Investigational Scan (Me-4FDG PET/CT) for the Detection of Sodium-Glucose Transport for Early Diagnosis of Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: LUNGevity Foundation (Other); American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-000027; NCI-2022-06770 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2022-09-12; First posted 2022-09-28 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-09

CONDITIONS: Lung Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — methyl-4-fluoro-4-deoxyglucose; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (Me-4FDG PET/CT) (Experimental): Patients receive Me-4FDG tracer IV and then undergo PET/CT over 15 minutes.
  Interventions: Drug: Alpha-methyl-4-deoxy-4-[(18)F]fluoro-D-glucopyranoside; Procedure: Computed Tomography; Other: Laboratory Biomarker Analysis; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: Alpha-methyl-4-deoxy-4-[(18)F]fluoro-D-glucopyranoside — Given IV
  Other Names: a-methyl-4[18F]-4-deoxy-D-glucopyranoside; Alpha-methyl-4-[F-18]-fluoro-4-deoxy-d-glucopyranoside; Me-4(18F)DG; Me-4FDG; Me4FDG; METHYL 4-DEOXY-4-FLUORO-.ALPHA.-D-GLUCOPYRANOSIDE. F-18
Procedure: Computed Tomography — Undergo PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized Tomography; CT; CT Scan; tomography
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging

SUMMARY:
The phase I/II trial assess the safety and efficacy of a new positron emission tomography (PET) test for early diagnosis of lung cancer. This study uses PET and Me-4FDG new glucose tracer (alpha-methyl-4-deoxy-4-[(18)F]fluoro-D-glucopyranoside) designed specifically to determine glucose update into cells in the body. PET is a non-invasive imaging method used to detect cancer in patient. Me4FDG is a radioactive glucose tracer used in PET to locate cells in the body taking up glucose by SGLT2. SLGT2 is a sodium glucose transport protein that accumulates glucose in some cells, e.g. kidney cells and tumors. This study may help researcher determine how effective PET with ME4FDG tracer works in detecting lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Assess the safety and efficacy of alpha-methyl-4-deoxy-4-[(18)F]fluoro-D-glucopyranoside (Me-4FDG) for early diagnosis of lung cancer.

SECONDARY OBJECTIVE:

I. Evaluate the correlation of Me-4FDG positivity with histopathological features of the disease (tumor grade, expression of sodium-glucose cotransporter-2 inhibitors.(SGLT2).

OUTLINE:

Patients receive Me-4FDG tracer intravenously (IV) and then undergo PET/CT over 15 minutes.

After completion of study , patients are followed up at 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Lung nodule >= 1 cm visualized by CT imaging
* CANCER ARM: Pathologically confirmed lung adenocarcinoma. For patients who are surgical candidates, the pathologic report on the surgical specimen will confirm the diagnosis. For patients who are not surgical candidates, the enrollment will be contingent upon a pathologic diagnosis of lung cancer obtained by needle biopsy
* BENIGN ARM: Lung nodules considered to be clinically benign, according to the Guidelines for Management of Incidental Pulmonary Nodules from the Fleischner Society. Will consider "benign" the nodules with a lung-RADS score of 1-3

Exclusion Criteria:

* Pregnancy
* Diagnosis of diabetes
* Current treatment with SGLT2 inhibitors or metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-19 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of Alpha-methyl-4-deoxy-4-[(18)F]fluoro-D-glucopyranoside (Me-4FDG) positron-emission tomography (PET) scans | within one month of surgery or biopsy
  Will be determined by calculating the standardized uptake value (SUV) in the lesions and the contrast to noise ratio (CNR) relative to an area of normal lung surrounding the lesion, and evaluated by assessing the percentage of patients with a pathologic diagnosis of lung cancer that results positive at Me-4FDG PET scans.
Specificity of Me-4FDG for lung cancer | within one week of experimental PET/CT scan
  Will be estimated by the percentage of Me-4FDG negativity in lung nodules that have been determined radiologically and/or clinically to be benign with a lung-RAD (Lung Imaging Reporting and Data System), score 1-3.
Optimal combination of sensitivity and specificity | within one week of experimental PET/CT scan
  Will combine SUV and CNR cut-points that yield the optimal combination of sensitivity (positivity within the adenocarcinoma group) and specificity (negativity with the benign group). Optimality will be based on the cut-points that maximize the Youden index (sum of the sensitivity plus specificity). Based on the combined cut point, will construct 95% confidence intervals for the sensitivity and specificity.
Incidence of adverse events of Me-4FDG | From baseline to one week after Me-4FDG administration
  Will tabulate the number of adverse events (AEs) and the severity of adverse events (SAEs) for the overall population as well as within subjects.
Efficacy of Me-4FDG in diagnosing lung cancer | within one week of the experimental PET/CT scan
  Will be evaluated by measuring the percentage of test positivity in patients with a pathological diagnosis of lung cancer.

SECONDARY OUTCOMES:
Correlation of Me-4FDG positivity with histopathological features (tumor grade) | within one month of surgery or biopsy
  Ordinal logistic regression will be used to assess the correlation between Me-4FDG uptake and tumor grade.
Correlation of Me-4FDG positivity with histopathological features (expression of SGLT2) | within two months of surgery or biopsy
  Will be evaluated experimentally with validated specific antibodies.

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Scafoglio, MD, PhD, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- Yesenia Calzada, Los Angeles, California, United States